CLINICAL TRIAL: NCT03491774
Title: Montessori Intervention for Individuals With Dementia: A Feasibility Study
Brief Title: Montessori Intervention for Individuals With Dementia: A Feasibility Study From Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PILL-Montessori Dementia
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Dementia; Memory Impairment
Keywords: memory impairment, montessori intervention, neurocognitive disorder
MeSH Terms: conditions — Dementia; Memory Disorders; Neurocognitive Disorders

STUDY DESIGN:
Intervention Model Description: It's a single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Montessori Intervention (Experimental): Participants will receive Montessori intervention for three months,twice weekly sessions over the period of three months.
  Interventions: Behavioral: Montessori Intervention

INTERVENTIONS:
Behavioral: Montessori Intervention — The Montessori method is a system of teaching developed by Maria Montessori based on principles to promote learning and independence in children. In the context of dementia care, this method has been tried in research settings in older people and was found to be effective in improving certain behavioral outcomes such as eating behaviors, agitation, and mood. The intervention is based on designing and offering activities that take into consideration the interests, needs, past experiences and preferences of participants. Importantly, participants demonstrating positive engagement with the intervention, suggesting that this may be a promising form of support to investigate and develop further for the care of people with dementia.

SUMMARY:
The study has both quantitative and qualitative components.

The objective of the quantitative study is:

1. To culturally adapt and refine Montessori activities for people living with dementia in Pakistan.
2. To determine the feasibility and acceptability of culturally-adapted group based Montessori intervention for people with dementia in Pakistan.
3. To build capacity and capability in dementia research (researcher training)

The objective of the qualitative study is:

To explore views on perceived effectiveness and sustainability of the study.

DETAILED DESCRIPTION:
Pakistan is the sixth most populous country in the world. Mental health services are limited in Pakistan particularly older adults mental health services are almost nonexistent. According to a recent report in Pakistan currently 8 million people are of age 65 and above who have long term physical and psychological health conditions. This is a tough challenge for the country due to its poor economic condition.Hence, there is a need to develop programs that can help and improve the health-related quality of life of this population in low resource settings.We need to do a lot more work to address this issue.

One possible low-cost, accessible, non-pharmacological intervention for BPSD (Behavioral Psychiatric symptoms of dementia) is the Montessori approach which is evidence based.The aim of the proposed project is to explore the feasibility and acceptability of using the Montessori intervention for people with dementia in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Participants with the following characteristics will be invited to participate in the study;

  * Diagnosed with any type of dementia according to DSM V.
  * Montreal Cognitive Examination Scale with a cutoff score 10
  * Age 60 years or older
  * Residents of study catchment area
  * Able to communicate in Urdu or English
  * Not having any serious visual or hearing impairment
  * Capacity to consent to study participation
  * Willing to come to (care home, hospitals, research centre) for session.
  * Willing to participate in up to 60 minutes session of the intervention, twice a week.
  * Having a study partner (spouse or adult child caregiver) who agrees to participate in the study

Exclusion Criteria:

* Participants with the following characteristics will not be eligible for the study;

  * Advanced stage dementia
  * Participants diagnosed with severe mental or physical illness which, in the judgement of the PI, precludes them from safely participating in the study.
  * Unable to give consent to take part in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of undertaking a trial of the intervention, as determined by: | 3rd month (post intervention)
  Recruitment and attrition rates

SECONDARY OUTCOMES:
Therapy logs | 3rd month (post intervention)
  Acceptability and tolerability of the intervention
Montreal Cognitive Examination: | Changes from baseline to 3rd month
  It assesses different cognitive domains, attention and concentration, executive functions, memory, language, visuo constructional skills, conceptual thinking, calculation and orientation. Score >26 shows cognitive impairment.(Nasreddine et al., 2005)
Quality of life assessment in Dementia DEMQol | Changes from baseline to 3rd month outcome
  It's a 28 item self-report questionnaire for people with dementia. It inquires about feelings, memory, and everyday life of the people with dementia. Score ranges from 28-112 with four-point Likert scale (1 = a lot, 2 = quite a bit, 3 = a little, 4 = not at all) for responses. (Smith et al., 2005)
Geriatric Depression Scale | Changes from baseline to 3rd month outcome
  It comprises of 15 items on which a score of >5 is suggestive of depression and a score of greater than or equal to 10 is indicative of depression.(Almeida & Almeida, 1999)

CONTACTS AND LOCATIONS:
Locations (1):
- Darul Skoun (Older Adult care home), Karachi, Sindh, Pakistan